CLINICAL TRIAL: NCT06611384
Title: Prevalence of Arrhythmias in Hemorrhagic Myocardial Infarction During the Acute Post-PCI Phase
Brief Title: Arrhythmias in Hemorrhagic Myocardial Infarction During the Acute Post-PCI Phase
Acronym: MIRON-RHYTHM
Status: Completed | Type: Observational
Sponsor: Rohan Dharmakumar (Other)
Responsible Party: Sponsor-Investigator, Rohan Dharmakumar, Executive Director, Krannert Cardiovascular Research Center, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 19978f
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Hemorrhagic Myocardial Infarction; CCS-AMI Reperfusion Injury; Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevalence of Arrhythmias in Hemorrhagic Myocardial Infarction During the Acute Post-PCI Phase

ELIGIBILITY:
1. Age 18-85 years
2. Index STEMI
3. Coronary angiogram with Primary coronary intervention
4. No contraindications for Cardiac MRI

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acute MI with Primary PCI
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Ventricular Arrhytmia | 24 hours
  Prevalence of Premature Ventricular Contractions (PVCs), Non-Sustained Ventricular Tachycardia (NSVT), and Ventricular Tachycardia/Ventricular Fibrillation (VT/VF) detected by post-PCI Holter monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Dharmakumar, PhD, Study Director — Indiana University School of Medicine; Keyur P Vora, MD MS FACC, Principal Investigator — Indiana University School of Medicine
Locations (2):
- IU School of Medicine/ IUHealth, Krannert Cardiovascular Research Center, Indianapolis, Indiana, United States
- Synergy Cardiovascular Research Center, Rajkot, India

IPD SHARING:
Plan to Share IPD: No